CLINICAL TRIAL: NCT05799183
Title: A Bioequivalence Study of SHR-1210 in Healthy Subjects
Brief Title: A SHR-1210 BE Study on Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's R&D Strategy adjusted
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SHR-1210-I-105
Record Dates: First submitted 2023-03-13; First posted 2023-04-05 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2023-09

CONDITIONS: Advanced Tumors
MeSH Terms: interventions — camrelizumab

STUDY DESIGN:
Intervention Model Description: This study is divided into two parts: pre-test and formal test. Each experiment will have two independent cohorts of subjects who will receive the treatment(SHR-1210 before process changes and SHR-1210 after process changes，respectively), and each cohort will be followed by 192 hours of blood sampling for pharmacokinetic assessments, with safety and tolerability.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pre-test: ARM A (Experimental): SHR-1210 before process changes 20 mg
  Interventions: Drug: SHR-1210
- Pre-test: ARM B (Experimental): SHR-1210 after process changes 20 mg
  Interventions: Drug: SHR-1210
- Formal Test: ARM A (Experimental): SHR-1210 before process changes 20 mg
  Interventions: Drug: SHR-1210
- Formal Test: ARM B (Experimental): SHR-1210 after process changes 20 mg
  Interventions: Drug: SHR-1210

INTERVENTIONS:
Drug: SHR-1210 — Subjects will receive treatment SHR-1210 before process changes 20 mg
  Arms: Formal Test: ARM A; Pre-test: ARM A
Drug: SHR-1210 — Subjects will receive treatment SHR-1210 after process changes 20 mg
  Arms: Formal Test: ARM B; Pre-test: ARM B

SUMMARY:
The purpose of this study is to assess the bioequivalence of SHR-1210 before and after process changes.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects aged ≥ 18;
2. Weigh at least 50 kg, and have a body mass index (BMI) ≥ 19 and ≤28 kg/m2;
3. Subjects agree to use reliable contraceptive measures (e.g., abstinence, sterilization, contraceptives, injectable contraceptives methylprogesterone or subcutaneous implantation in the duration of the study and for 4 months after the study drug infusion);
4. Sign the informed consent before the trial, and fully understand the content, process and possible adverse reactions of the trial. Must be able to communicate with the investigator, understand and comply with all study requirements.

Exclusion Criteria:

1. Those with a history of chronic liver, kidney, cardiovascular, neurological/psychiatric, digestive tract, respiratory, urinary, endocrine and other systemic diseases;
2. Those with a history of autoimmune diseases;
3. Regular drinkers in the 6 months prior to the trial had an average daily alcohol intake of more than 15 g (equivalent to 145 mL of wine, 450 mL of beer, or 43 mL of liquor with 40% alcohol content);
4. Those who are suspected or confirmed to be allergic or have had serious drug or food allergic reactions in the past, have a clear history of allergies and/or are allergic to the research drug or its ingredients;
5. Have used any drug (including Chinese medicine and vitamins) within 2 weeks before screening, or the last dose is less than 5 half-lives of the drug from the test administration date, whichever is longer;
6. Have used of anti-PD-1/PD-L1 drugs;
7. Those who have participated in other interventional clinical trials within 3 months before screening;
8. ≥400 ml of blood loss, blood donation or receiving any blood product transfusion within 3 months before screening;
9. Those who have undergone major surgery or hospitalized for illness within 3 months before screening;
10. Those who have received live vaccines within 6 months prior to screening, or who are expected to receive live vaccines during the study period;
11. Those with a history of drug abuse or positive drug screening results within 12 months prior to screening;
12. Those who have abnormalities in vital signs, physical examination, and laboratory tests during the screening period and are judged to be clinically significant by the study physician (Note: If there is an abnormality and the study doctor judges that it has clinical significance, if it is within the normal range after re-examination, it can also be enrolled);
13. There are abnormalities in the ECG during the screening period (such as QTcF≥ 450ms, shortened or prolonged PR interval, second-degree and third-degree atrioventricular block, pre-excitation syndrome, etc.) and are judged by the study doctor to have clinical significance;
14. Chest x-ray (positive and lateral position) or lung CT during the screening period is abnormal and judged by the study doctor to be clinically significant;
15. History of needle sickness and blood sickness; or those with poor vascular conditions, unable to retain implanted needles or unable to tolerate venipuncture blood collection;
16. Those that the investigator believes are not suitable to participate in this clinical trial for other reasons.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-07-04 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
Pre-test: Incidence and severity of AE/SAE/AESI (rated based on CTCAE v5.0) | Day-1 to Day 46
Formal Test: Pharmacokinetics parameters of SHR-1210 before and after process changes in the fed state: AUC0-inf | Based on pre-dose, 0.25-192 hours post-dose sampling times on Day 1 ~ Day 4 and Day 6 ~ Day 9
Formal Test: Pharmacokinetics parameters of SHR-1210 before and after process changes in the fed state: the geometric mean ration | Based on pre-dose, 0.25-192 hours post-dose sampling times on Day 1 ~ Day 4 and Day 6 ~ Day 9
Formal Test: Pharmacokinetics parameters of SHR-1210 before and after process changes in the fed state: 90% confidence interval (90% CI) of AUC0-inf | Based on pre-dose, 0.25-192 hours post-dose sampling times on Day 1 ~ Day 4 and Day 6 ~ Day 9

SECONDARY OUTCOMES:
Pre-test: Inter-individual coefficient of variation (CV) of the AUC0-inf of SHR-1210 | Based on pre-dose, 0.25-192 hours post-dose sampling times on Day 1 ~ Day 4 and Day 6 ~ Day 9
Formal Test: Other Pharmacokinetics parameters of SHR-1210 before and after process changes in the fed state: Cmax | Based on pre-dose, 0.25-192 hours post-dose sampling times on Day 1 ~ Day 4 and Day 6 ~ Day 9
Formal Test: Other Pharmacokinetics parameters of SHR-1210 before and after process changes in the fed state: AUC0-t | Based on pre-dose, 0.25-192 hours post-dose sampling times on Day 1 ~ Day 4 and Day 6 ~ Day 9
Formal Test: Other Pharmacokinetics parameters of SHR-1210 before and after process changes in the fed state: Tmax | Based on pre-dose, 0.25-192 hours post-dose sampling times on Day 1 ~ Day 4 and Day 6 ~ Day 9
Formal Test: Other Pharmacokinetics parameters of SHR-1210 before and after process changes in the fed state: t1/2 | Based on pre-dose, 0.25-192 hours post-dose sampling times on Day 1 ~ Day 4 and Day 6 ~ Day 9
Formal Test: Other Pharmacokinetics parameters of SHR-1210 before and after process changes in the fed state: CL | Based on pre-dose, 0.25-192 hours post-dose sampling times on Day 1 ~ Day 4 and Day 6 ~ Day 9
Formal Test: Other Pharmacokinetics parameters of SHR-1210 before and after process changes in the fed state: Vss | Based on pre-dose, 0.25-192 hours post-dose sampling times on Day 1 ~ Day 4 and Day 6 ~ Day 9
Formal Test: The incidence of anti-drug antibody (ADA) and neutralizing antibody (Nab) for SHR-1210 | Based on sampling times pre-dose on Day1, post-dose on Day 9 and Day 16
Formal Test: Incidence and severity of adverse events (rated based on CTCAE 5.0） | Day-1, Day 1 to Day 46±7

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided